CLINICAL TRIAL: NCT02723864
Title: Phase I Study of Veliparib (ABT-888), an Oral PARP Inhibitor, and VX-970, an ATR Inhibitor in Combination With Cisplatin in Patients With Refractory Solid Tumors
Brief Title: Veliparib (ABT-888), an Oral PARP Inhibitor, and VX-970, an ATR Inhibitor, in Combination With Cisplatin in People With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160087; 16-C-0087
Record Dates: First submitted 2016-03-30; First posted 2016-03-31 (Estimated); Results first posted 2022-01-10 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Neoplasms
Keywords: Pharmacodynamic; DNA Damage Repair; BRCA Null; Apoptosis; Combination Therapy
MeSH Terms: conditions — Neoplasms | interventions — veliparib; berzosertib; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- M6620 (VX-970) (Experimental): M6620 will be administered intravenous (IV) on Days 2 and 9 of each 21-day cycle; Veliparib will be administered orally twice a day (BID) Days 1-3 and 8-10 of each cycle; Cisplatin will be administered at 40 mg/m^2 IV Day 1 (and Day 8 from dose level 3 onwards) of each cycle
  Interventions: Drug: Veliparib + VX-970 + Cisplatin

INTERVENTIONS:
Drug: Veliparib + VX-970 + Cisplatin — Ataxia-telangiectasia-related (ATR) protein kinase is central to the deoxyribonucleic acid (DNA) damage response and homologous recombination, activating a series of phosphorylation cascades, culminating in cell cycle arrest to allow time for DNA repair. Poly (ADP-ribose) polymerase (PARP) plays a pivotal role in base-excision repair of single strand breaks formed either due to direct genotoxic stress or during the processing of double strand breaks. Preclinical studies show ATR inhibitor M6620 (VX-970) synergizes with cisplatin to induce DNA damage and antitumor activity. The addition of PARP inhibitor veliparib with VX-970 allows for impairment of DNA repair, induction of a breast cancer gene (BRCA) null phenotype, and potentiation of the antitumor activity of cisplatin.
  Other Names: ABT-888 + M6620 (berzosertib) + Cisplatinum

SUMMARY:
Background:

The drug cisplatin treats certain cancers when given with other chemotherapy drugs. Researchers think combining cisplatin with 2 other drugs could block proteins that support cancer cell growth. The other drugs are ABT-888 (veliparib) and M6620 (VX-970). They want to test if this drug combination slows the growth of cancer and is safe.

Objectives:

To test the safety and tolerability of VX-970 and veliparib combined with cisplatin in people with advanced refractory solid tumors. To determine the maximum tolerated dose of these drugs.

Eligibility:

People ages 18 and older with:

* Solid tumors that have progressed after treatment or for which no treatment exists
* Normal organ and marrow function

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Computed tomography (CT) scan or magnetic resonance imaging (MRI)
* Blood and urine tests

Participants will get the study drugs in 3-week cycles:

* Cisplatin in a vein on 1 or 2 days
* VX-970 in a vein on 2 days
* Veliparib by mouth twice a day on 6 days

In each cycle, participants will have 5 physical exams and blood tests 5 times.

In some cycles, participants will have CT scans or MRIs.

In cycle 1, participants may have 2 tumor biopsies. A small piece of tissue is removed by needle.

Participants will keep a study diary. They will write when they take the drugs and if they have side effects.

Participants will stay in the study as long as they tolerate the drugs and their tumors are not getting worse.

Participants will have a phone call about a month after their last dose.

DETAILED DESCRIPTION:
Background:

* Ataxia-telangiectasia-related (ATR) protein kinase is central to the deoxyribonucleic acid (DNA) damage response and homologous recombination, activating a series of phosphorylation cascades, culminating in cell cycle arrest to allow time for deoxyribonucleic acid (DNA) repair. ATR additionally facilitates homologous recombination repair through modulation of the p53-replication protein A (p53-RPA) complex bound to single-stranded deoxyribonucleic acid (ssDNA) during the DNA repair process.
* Poly (ADP-ribose) polymerase-1 (PARP-1) plays a pivotal role in base-excision repair of single strand breaks formed either due to direct genotoxic stress or during the processing of double strand breaks. PARP also plays a role in alternative end joining, which may contribute to combination activity. PARP-1 binding to sites of DNA damage results in activation of its catalytic activity and generation of chains of poly (ADP-ribosyl)ated polymers, which serve as docking sites for recruitment of DNA repair proteins.
* Veliparib (ABT-888) is a potent PARP 1/2 inhibitor with clinical evidence of potentiation of antitumor activity in combination with cisplatin in breast cancer gene (BRCA) mutation carriers and patients with sporadic triple-negative breast cancer.
* M6620 (VX-970) is a potent ATR inhibitor, with half maximal inhibitory concentration (IC(50) of 20 nanomolar and antitumor activity across a broad range of cell lines in combination with DNA damaging agents. Preclinical studies show M6620 (VX-970) synergizes with cisplatin to induce DNA damage and antitumor activity. The addition of PARP inhibitor veliparib with ATR inhibitor M6620 (VX-970) allows for impairment of DNA repair, the induction of a BRCA null phenotype, and potentiation of the antitumor activity of cisplatin.

Primary Objective:

-To establish the safety, tolerability, and the maximum tolerated dose (MTD) of the combination of M6620 (VX-970) and veliparib in combination with cisplatin in patients with advanced refractory solid tumors

Secondary Objectives:

* To assess the effect of the combination of M6620 (VX-970), veliparib, and cisplatin on markers of DNA damage and apoptosis
* To assess antitumor activity of the combination

Exploratory Objective:

-To investigate tumor genomic alterations potentially associated with acquired resistance to the combination of M6620 (VX-970), veliparib, and cisplatin

Eligibility:

* Patients must have histologically confirmed solid tumors for which all standard therapy known to prolong survival has failed in the metastatic setting, or for which standard therapies do not exist
* Patients must have had no major surgery, radiation, or chemotherapy within 3 weeks prior to entering the study
* Patients must have adequate organ function

Study Design:

* Initially, M6620 (VX-970) will be administered intravenously on Days 2 and 9 of each 21-day cycle. Veliparib will be administered orally twice a day (every (q)12 hours +/- 1 hour) for Days 1-3 and 8-10 of each 21-day cycle. Cisplatin will be administered at 40 mg/m^2 intravenously on Day 1 (and Day 8 from dose level 3 (DL3) onwards) of each 21-day cycle.
* As of Amendment I (12/7/2017), patients who have been on study for at least 6 cycles may have cisplatin administration held or discontinued at the discretion of the Principal Investigator (PI), Dr. Chen, in recognition of the cumulative neurotoxicity seen with cisplatin treatment. If cisplatin is not administered during a cycle M6620 (VX-970) will be administered on Days 1 and 8 of that cycle.
* The escalation portion of the trial will follow a standard 3+3 design, whereby patients will be dose escalated in cohorts of 3 until dose-limiting toxicity is observed
* Once the maximum tolerated dose (MTD) is established, up to 15 additional patients will be enrolled to an expansion phase at the MTD. Mandatory tumor biopsies will be obtained in the expansion phase to assess pharmacodynamic (PD) endpoints

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed solid tumors for which standard therapy known to prolong survival has failed in the metastatic setting or for which standard therapies do not exist.
* Tumor amenable to biopsy and willingness to undergo tumor biopsies before and after M6620 (VX-970) treatment during the expansion phase of the trial (biopsies optional during the escalation phase).
* Patients must have completed any chemotherapy, radiation therapy, surgery, or biologic therapy greater than or equal to 3 weeks (or greater than or equal to 5 half-lives, whichever is shorter) prior to entering the study. Patients must be greater than or equal to 2 weeks since any prior administration of a study drug in an exploratory investigational new drug (IND)/Phase 0 study and greater than or equal to 1 week since any palliative radiation therapy. Patients must have recovered to eligibility levels from prior toxicity or adverse events.
* Age greater than or equal to 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Life expectancy > 3 months.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/mcL
  * hemoglobin greater than or equal to 10 g/dL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin less than or equal to 1.5 X institutional upper limit of normal
  * Aspartate aminotransferase (AST) Serum glutamic oxaloacetic transaminase(SGOT)/alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase (SGPT) less than or equal to 1.5 X institutional upper limit of normal (OR < 3X upper limit of normal (ULN) in the setting of liver metastases)
  * creatinine less than or equal to 1.5X institutional upper limit of normal

OR

* creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal

  * The effects of M6620 (VX-970) and veliparib on the developing human fetus are unknown. For this reason and because cisplatin is known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after completing study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 6 months after completion of administration of study agents.
  * Human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with M6620 (VX-970). In addition, these subjects are at increased risk of lethal infections when treated with marrow-suppressive therapy.
  * Patients must be able to swallow whole tablets or capsules. Nasogastric or gastric (G)-tube administration is not allowed. Any gastrointestinal disease which would impair ability to swallow, retain, or absorb drug is not allowed.
  * Ability to understand and the willingness to sign a written informed consent document.
  * During the expansion phase of the protocol, patients must have disease amenable to biopsy and be willing to undergo pre- and post-treatment biopsies.
  * Patients must have greater than or equal to 10.0 g/dL hemoglobin (Hb) and no blood transfusion in the past 28 days to receive Veliparib.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Patients with known active brain metastases or carcinomatous meningitis are excluded from this clinical trial. Patients whose brain metastatic disease status has remained stable for greater than or equal to 4 weeks following treatment of brain metastases are eligible to participate at the discretion of the principal investigator.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active untreated infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients required to be on any of the concomitant medications are excluded.
* Pregnant women and women who are breastfeeding are excluded from this study because the effects of the study drugs on the developing fetus are unknown.
* Patients who have had prior platinum-based therapy who have > Grade 1 neurotoxicity or ototoxicity at the time of enrollment will not be permitted on study.
* Patients with a seizure history will not be permitted on protocol due to association of veliparib with seizure activity in animal toxicology studies at higher doses. Patients on anticonvulsant medications will not be permitted on study due to the potential to lower plasma levels of anticonvulsants and risk for seizure activity.
* Patients with treatment-related acute myeloid leukemia (AML) (t-AML)/Myelodysplastic syndromes (MDS), or with features suggestive of AML/MDS, or who have had prior allogeneic bone marrow transplant or double umbilical cord blood transplantation, should not receive Veliparib due to reports of MDS and leukemia secondary to oncology therapy on Cancer Therapy Evaluation Program (CTEP)-sponsored studies utilizing Veliparib.

INCLUSION of WOMEN and MINORITIES

Both men and women of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
We will share IPD (clinical data) during the study and indefinitely via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: During the study and indefinitely via subscription to Biomedical Translational Research Information System (BTRIS).
Access Criteria: IPD will be shared with NIH Intramural investigators who provide a methodologically sound proposal and whose proposed use of the data has been approved by the study PI, for the purpose of achieving the aims in the approved proposals. Proposals should be submitted via subscription to Biomedical Translational Research Information System (BTRIS).
URL: http://btris.nih.gov/

REFERENCES:
- [Background] Chen X, Wu Y, Dong H, Zhang CY, Zhang Y. Platinum-based agents for individualized cancer treatment. Curr Mol Med. 2013 Dec;13(10):1603-12. doi: 10.2174/1566524013666131111125515. PMID 24206132
- [Background] Huntoon CJ, Flatten KS, Wahner Hendrickson AE, Huehls AM, Sutor SL, Kaufmann SH, Karnitz LM. ATR inhibition broadly sensitizes ovarian cancer cells to chemotherapy independent of BRCA status. Cancer Res. 2013 Jun 15;73(12):3683-91. doi: 10.1158/0008-5472.CAN-13-0110. Epub 2013 Apr 2. PMID 23548269
- [Background] Donawho CK, Luo Y, Luo Y, Penning TD, Bauch JL, Bouska JJ, Bontcheva-Diaz VD, Cox BF, DeWeese TL, Dillehay LE, Ferguson DC, Ghoreishi-Haack NS, Grimm DR, Guan R, Han EK, Holley-Shanks RR, Hristov B, Idler KB, Jarvis K, Johnson EF, Kleinberg LR, Klinghofer V, Lasko LM, Liu X, Marsh KC, McGonigal TP, Meulbroek JA, Olson AM, Palma JP, Rodriguez LE, Shi Y, Stavropoulos JA, Tsurutani AC, Zhu GD, Rosenberg SH, Giranda VL, Frost DJ. ABT-888, an orally active poly(ADP-ribose) polymerase inhibitor that potentiates DNA-damaging agents in preclinical tumor models. Clin Cancer Res. 2007 May 1;13(9):2728-37. doi: 10.1158/1078-0432.CCR-06-3039. PMID 17473206
- [Derived] O'Sullivan Coyne G, Do KT, Kummar S, Piha-Paul S, Rubinstein L, Kinders R, Parchment RE, Wilsker D, Ferry-Galow K, Miller B, Takebe N, Juwara L, Ong MJ, Bruns A, Hogu M, Naqash AR, Mittra A, Voth AR, Doroshow JH, Chen AP. Safety and Tolerability of Berzosertib, an Ataxia-Telangiectasia-Related Inhibitor, and Veliparib, an Oral Poly (ADP-ribose) Polymerase Inhibitor, in Combination With Cisplatin in Patients With Refractory Solid Tumors. JCO Precis Oncol. 2025 Jul;9:e2500055. doi: 10.1200/PO-25-00055. Epub 2025 Jul 16. PMID 40669022
- [Derived] Smith G, Alholm Z, Coleman RL, Monk BJ. DNA Damage Repair Inhibitors-Combination Therapies. Cancer J. 2021 Nov-Dec 01;27(6):501-505. doi: 10.1097/PPO.0000000000000561. PMID 34904813
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0087.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: DL 1: ABT-888 100 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 90 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr day 1 (optional after 6 cycles)
- Dose Level 2: DL 2: ABT-888 100 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 140 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr day 1 (optional after 6 cycles)
- Dose Level 3: DL 3: ABT-888 100 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 120 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr days 1 & 8 (optional after 6 cycles)
- Dose Level 4: DL 4: ABT-888 100 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 210 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr days 1 & 8 (optional after 6 cycles)
- Dose Level 5: DL 5: ABT-888 150 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 210 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr days 1 & 8 (optional after 6 cycles)
- Dose Level 6: DL 6: ABT-888 200 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 210 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr days 1 & 8 (optional after 6 cycles)
- Dose Level 7: DL 7: ABT-888 300 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 210 mg/m^2 IV over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 intravenous (IV) over 1hr days 1 & 8 (optional after 6 cycles)
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Dose Level 7
Started | 3 | 3 | 6 | 7 | 3 | 25 | 6
Completed | 2 | 2 | 5 | 7 | 2 | 14 | 4
Not Completed | 1 | 1 | 1 | 0 | 1 | 11 | 2
Not completed — Refused further treatment | 1 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Exceed treatment hold time | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical progression | 0 | 0 | 1 | 0 | 0 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Changes in patient condition | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Patient choice | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Started new treatment | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Switched to alternative treatment | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Late determination of ineligibility | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Dose Level 7 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 25 | 6 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 6 | 5 | 3 | 20 | 6 | 44
  >=65 years | 1 | 1 | 0 | 2 | 0 | 5 | 0 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.67 (7.64) | 51 (15.39) | 54.83 (10.65) | 57.86 (13.21) | 58 (5.57) | 53.4 (14.28) | 44.83 (14.3) | 53.6 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 6 | 5 | 1 | 9 | 4 | 27
  Male | 3 | 1 | 0 | 2 | 2 | 16 | 2 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
  Not Hispanic or Latino | 3 | 3 | 6 | 7 | 2 | 21 | 6 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 3 | 1 | 3 | 0 | 8
  White | 3 | 3 | 5 | 4 | 2 | 19 | 6 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 7 | 3 | 25 | 6 | 53
Eastern Cooperative Oncology Performance Status (ECOG) [Count of Participants; unit: Participants] — ECOG performance status 0 is fully active. ECOG performance status 1 is symptoms but ambulatory. ECOG performance status 2 is in bed <50% of the time.
  Participants
    ECOG 0 | 0 | 0 | 2 | 0 | 0 | 5 | 2 | 9
    ECOG 1 | 2 | 3 | 4 | 7 | 3 | 19 | 4 | 42
    ECOG 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Diagnosis: Tumor Type [Count of Participants; unit: Participants]
  Lung cancer | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Ovarian cancer | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 6
  Liver cancer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Uterine cancer | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Pancreatic cancer | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 5
  Peritoneal cancer | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Breast cancer | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3
  Colon cancer | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3
  Esophageal cancer | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Other | 1 | 2 | 1 | 5 | 3 | 14 | 4 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Worst Grade 2 or Higher Adverse Events Occurring in >5% of Participants at Least Possibly Related to Study Drugs
Description: Adverse events were assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 2 is moderate, Grade 3 is severe or medically significant but not immediately life threatening, and Grade 4 is life threatening.
Time Frame: Cycle 1 (i.e., one cycle = 21 days)
Measure: Count of Participants; unit: Participants
Groups:
- Grade 2 Adverse Events - Dose Level 1; Grade 3 Adverse Events - Dose Level 1; Grade 4 Adverse Events - Dose Level 1: DL 1: ABT-888 100 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 90 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr day 1 (optional after 6 cycles)
- Grade 2 Adverse Events - Dose Level 2; Grade 3 Adverse Events - Dose Level 2; Grade 4 Adverse Events - Dose Level 2: DL 2: ABT-888 100 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 140 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr day 1 (optional after 6 cycles)
- Grade 2 Adverse Events - Dose Level 3; Grade 3 Adverse Events - Dose Level 3; Grade 4 Adverse Events - Dose Level 3: DL 3: ABT-888 100 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 120 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr days 1 & 8 (optional after 6 cycles)
- Grade 2 Adverse Events - Dose Level 4; Grade 3 Adverse Events - Dose Level 4; Grade 4 Adverse Events - Dose Level 4: DL 4: ABT-888 100 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 210 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr days 1 & 8 (optional after 6 cycles)
- Grade 2 Adverse Events - Dose Level 5; Grade 3 Adverse Events - Dose Level 5; Grade 4 Adverse Events - Dose Level 5: DL 5: ABT-888 150 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 210 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr days 1 & 8 (optional after 6 cycles)
- Grade 2 Adverse Events - Dose Level 6; Grade 3 Adverse Events - Dose Level 6; Grade 4 Adverse Events - Dose Level 6: DL 6: ABT-888 200 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 210 mg/m^2 intravenous (IV) over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 IV over 1hr days 1 & 8 (optional after 6 cycles)
- Grade 2 Adverse Events - Dose Level 7; Grade 3 Adverse Events - Dose Level 7; Grade 4 Adverse Events - Dose Level 7: DL 7: ABT-888 300 mg by mouth (PO) every (Q)12 hours on days 1-3 & 8-10, VX-970 210 mg/m^2 IV over 1 hour days 2 & 9, Cisplatin 40 mg/m^2 intravenous (IV) over 1hr days 1 & 8 (optional after 6 cycles)
Arm/Group | Grade 2 Adverse Events - Dose Level 1 | Grade 3 Adverse Events - Dose Level 1 | Grade 4 Adverse Events - Dose Level 1 | Grade 2 Adverse Events - Dose Level 2 | Grade 3 Adverse Events - Dose Level 2 | Grade 4 Adverse Events - Dose Level 2 | Grade 2 Adverse Events - Dose Level 3 | Grade 3 Adverse Events - Dose Level 3 | Grade 4 Adverse Events - Dose Level 3 | Grade 2 Adverse Events - Dose Level 4 | Grade 3 Adverse Events - Dose Level 4 | Grade 4 Adverse Events - Dose Level 4 | Grade 2 Adverse Events - Dose Level 5 | Grade 3 Adverse Events - Dose Level 5 | Grade 4 Adverse Events - Dose Level 5 | Grade 2 Adverse Events - Dose Level 6 | Grade 3 Adverse Events - Dose Level 6 | Grade 4 Adverse Events - Dose Level 6 | Grade 2 Adverse Events - Dose Level 7 | Grade 3 Adverse Events - Dose Level 7 | Grade 4 Adverse Events - Dose Level 7
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 7 | 7 | 7 | 3 | 3 | 3 | 25 | 25 | 25 | 6 | 6 | 6
Participants
  Alkaline phosphatase increased | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 3 | 3 | 0 | 0 | 3 | 0 | 6 | 10 | 1 | 1 | 2 | 0
  Creatinine increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Fatigue | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0
  Hypertension | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 0 | 1 | 1 | 0
  Hypomagnesemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  Hyponatremia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypophosphatemia | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  Infusion related reaction | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
  Lymphocyte count decreased | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 1 | 1 | 0 | 0
  Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 3 | 1
  Peripheral sensory neuropathy | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 1 | 0 | 2 | 0 | 2 | 4 | 3 | 1 | 1 | 1
  Proteinuria | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Thromboembolic event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0
  White blood cell decreased | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 4 | 4 | 1 | 1 | 2 | 0

2. Secondary Outcome: Number of Participants With RAD51 Recombinase (Rad51), Phosphorylated Histone H2AX (γH2AX), Phosphorylated at Serine 343 (pS343)-Nibrin (Nbs1), and Phosphorylated KRAB-associated Protein 1 (pKAP-1) Induced After Treatment
Description: Biopsies were collected at Cycle 1 Day 1, and Cycle 1 Day 9 and markers Rad51, γH2AX, pS343-Nbs1, and pKAP-1 were measured for deoxyribonucleic acid (DNA) damage and apoptosis by immunofluorescence assays (IFA).
Time Frame: Cycle 1 Day 1, and Cycle 1 Day 9 (i.e., one cycle = 21 days)
Population: These measurements were only carried out on the subset (7/25) of DL6 participants from whom evaluable C1D1 and C1D9 biopsies were collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Dose Level 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 0
Participants
  Rad51 induced after veliparib and cisplatin treatment on Cycle 1, Day 1 |  |  |  |  |  | 5 |
  Rad51 induced after veliparib, cisplatin and M6620 treatment on Cycle 1, Day 9 |  |  |  |  |  | 5 |
  γH2AX induced after veliparib and cisplatin treatment on Cycle 1, Day 1 |  |  |  |  |  | 0 |
  γH2AX induced after veliparib, cisplatin and M6620 treatment on Cycle 1, Day 9 |  |  |  |  |  | 0 |
  pS343-Nbs1 induced after veliparib and cisplatin treatment on Cycle 1, Day 1 |  |  |  |  |  | 1 |
  pS343-Nbs1 induced after veliparib, cisplatin and M6620 treatment on Cycle 1, Day 9 |  |  |  |  |  | 0 |
  pKap1 induced after veliparib and cisplatin treatment on Cycle 1, Day 1 |  |  |  |  |  | 0 |
  pKap1 induced after veliparib, cisplatin and M6620 treatment on Cycle 1, Day 9 |  |  |  |  |  | 0 |

3. Secondary Outcome: Number of Participants With a Best Response to the Antitumor Activity of Veliparib (ABT-888), an Oral PARP Inhibitor, and VX-970, an ATR Inhibitor, in Combination With Cisplatin
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, and the appearance of one or more new lesions. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: 4 cycles (i.e., one cycle = 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Dose Level 7
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 25 | 6
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 2 | 0 | 0 | 3 | 0
  Stable Disease | 1 | 2 | 3 | 4 | 3 | 10 | 3
  Progressive Disease | 2 | 1 | 1 | 3 | 0 | 5 | 3
  Not Evaluable for Response | 0 | 0 | 0 | 0 | 0 | 7 | 0

4. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 6 months and 20 days, 3 months and 17 days, 24 months and 13 days, 9 months and 8 days, 5 months and 18 days, 35 months and 20 days, and 5 months and 22 days for each Arm/Group respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Dose Level 7
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 25 | 6
Participants | 3 | 3 | 6 | 7 | 3 | 25 | 6

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 6 months and 20 days, 3 months and 17 days, 24 months and 13 days, 9 months and 8 days, 5 months and 18 days, 35 months and 20 days, and 5 months and 22 days for each Arm/Group respectively.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Dose Level 7
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/7 | 0/3 | 1/25 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/6 | 2/7 | 1/3 | 14/25 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 7/7 | 3/3 | 25/25 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=6) | Dose Level 4 (N=7) | Dose Level 5 (N=3) | Dose Level 6 (N=25) | Dose Level 7 (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=6) | Dose Level 4 (N=7) | Dose Level 5 (N=3) | Dose Level 6 (N=25) | Dose Level 7 (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 5 (7) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 3 (5) | 1 (5) | 0 (0) | 4 (4) | 2 (3)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 3 (6) | 2 (7) | 1 (1) | 3 (4) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (9) | 3 (4) | 6 (57) | 6 (35) | 3 (21) | 19 (81) | 4 (19)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (6) | 2 (3) | 2 (2) | 9 (11) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (3) | 2 (5) | 1 (2) | 7 (7) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (2) | 2 (5) | 3 (4) | 0 (0) | 11 (15) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 4 (6) | 3 (5) | 0 (0) | 6 (18) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (6) | 3 (3) | 1 (2) | 11 (24) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 2 (2) | 1 (2) | 1 (2) | 0 (0) | 4 (5) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (4) | 5 (6) | 0 (0) | 8 (10) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 4 (10) | 1 (1) | 0 (0) | 5 (7) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Eye disorders - Other, Sty (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Fatigue (General disorders) | 3 (5) | 3 (5) | 4 (6) | 4 (7) | 2 (4) | 13 (16) | 5 (7)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Gastrointestinal disorders - Other, Cramping abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 3 (4) | 3 (3) | 1 (1) | 4 (5) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (3) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 1 (1) | 2 (6) | 1 (12) | 14 (25) | 3 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (6) | 2 (4) | 4 (27) | 2 (7) | 0 (0) | 13 (54) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 1 (4) | 1 (2) | 2 (4) | 8 (23) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 5 (12) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 5 (10) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4) | 2 (5) | 4 (10) | 3 (6) | 1 (1) | 8 (32) | 3 (6)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4) | 2 (4) | 3 (8) | 2 (8) | 2 (4) | 11 (24) | 4 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (8) | 2 (3) | 3 (7) | 2 (7) | 1 (1) | 6 (13) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, c diff infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (3)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (4) | 3 (3) | 1 (1) | 1 (2) | 1 (1) | 6 (8) | 1 (1)
Investigations - Other, hyponatremia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, LDH Inc (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (17) | 2 (10) | 2 (12) | 1 (7) | 1 (4) | 9 (74) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (2) | 3 (7) | 4 (4) | 1 (1) | 14 (17) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (2) | 2 (5) | 5 (15) | 4 (12) | 1 (2) | 7 (56) | 5 (12)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Phlebitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (6) | 3 (5) | 4 (13) | 7 (27) | 2 (13) | 17 (62) | 5 (17)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal and urinary disorders - Other, dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, glucosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (20) | 1 (1) | 0 (0) | 11 (25) | 3 (4)
Skin and subcutaneous tissue disorders - Other, Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, chest redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, nail change (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (4) | 2 (2) | 0 (0) | 8 (14) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
White blood cell decreased (Investigations) | 1 (7) | 2 (8) | 2 (15) | 5 (20) | 2 (11) | 11 (81) | 4 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT02723864/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT02723864/ICF_001.pdf